CLINICAL TRIAL: NCT04213339
Title: Effectiveness of Kegal Exercises on Urinary Incontinence Impact in Geriatric Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zohra Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Suhail Karim, Assistant Professor, Riphah International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZIHS-Rwp/IRC/003
Record Dates: First submitted 2019-12-27; First posted 2019-12-30 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Urinary Incontinence in Geriatric Population

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kegal Exercises (Experimental)
  Interventions: Behavioral: Kegel Exercises
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Kegel Exercises — Kegel exercise group will get exercise within duration of 3 to 6 weeks based on age factor. Kegel exercise can be performed at any time and at any place without any restrictions.
  following steps will be followed by kegel exercises group members:
  1. Tighten and hold pelvic floor muscles for five seconds (count 1 one thousand, 2 one thousand, 3 one thousand, 4 one thousand, 5 one thousand).
  2. Relax pelvic muscles and perform 10 to 20 Kegel exercises three to four times each day.
  3. Squeeze the muscles in anus like holding a bowel movement focus penile area
  4. Relax the pelvic floor muscles after each attempt.
  5. Repeat this exercise 10 to 20 times.
  6. While performing Kegel exercises:
  Do not hold the breath. Do not push down. Squeeze the muscles together tightly and imagine, trying to lift this muscle up. Do not tighten the muscles in the stomach, buttocks, or thighs.
  While the control group did not participate in any kegel exercises
  Arms: Kegal Exercises

SUMMARY:
This research study was used to determine effectiveness of kegal exercise on urinary incontinence impact in geriatric incontinence. There were two groups, One group was experimental which was subjected to Kegel exercises while other was control group without any treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient 50 years of age and above.
* Geriatric population
* Male participant

Exclusion Criteria:

* Patient below 50 years of age.
* Patient with neurological problem.
* Uncooperative attitude
* Male patients with prostate problem & Female participants

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male old age geriatric population
Enrollment: 50 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Incontinence Impact | 6 to 8 weeks
  Incontinence impact questionnaire description:
  For each question, circle the response that best describes how much your activities, relationships, and feelings are being affected by urine leakage.
  Scoring: Items 1 and 2 = physical activity Items 3 and 4 = travel Item 5 = social/relationships Items 6 and 7 = emotional health
  Scoring. Item responses are assigned values of 0 for "not at all," 1 for "slightly," 2 for "moderately," and 3 for "greatly." The average score of items responded to is calculated. The average, which ranges from 0 to 3, is multiplied by 33 1/3 to put scores on a scale of 0 to 100.
  1. Ability to do household chores
  2. Physical recreation such as walking, swimming, or other exercise?
  3. Entertainment activities
  4. Ability to travel by car or bus more than 30 minutes from home.
  5. Participation in social activities outside your home
  6. Emotional health
  7. Feeling frustrated?

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Sikandar Bhutto, Rawalpindi, Pakistan